CLINICAL TRIAL: NCT04491851
Title: A Prospective Study to Evaluate the Impact of Different Peptides and Chelators on the Diagnostic Performance of PET/CT Using Gallium-68 Labeled Somatostatin Receptor Antagonists
Brief Title: Impact of Peptides and Chelators on Somatostatin Receptor Antagonists
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ANTANET
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Neuroendocrine Tumors
Keywords: somatostatin receptor antagonist; PET/CT
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into four arms:
  Arm A : 68Ga-NODAGA-LM3 and 68Ga-DOTA-LM3 Arm B : 68Ga-NODAGA-LM3 and 68Ga-NODAGA-JR11
Who Masked: Participant, Outcomes Assessor
Masking Description: The details of patient groups will be sealed in sequentially numbered, opaque, sealed envelopes generated by Xuezhu Wang from the nuclear medicine department, Peking Union Medical College Hospital, who will not participate in other parts of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM3 group (Experimental): In this arm, patients will undergo PET/CT using 68Ga-NODAGA-LM3 (40ug peptide/150-200MBq) and 68Ga-DOTA-LM3 (40ug peptide/150-200MBq) on two consecutive days. The scan will be acquired at 1hour post-injection.
  Interventions: Diagnostic Test: 68Ga-NODAGA-LM3 and 68Ga-DOTA-LM3 PET/CT
- NODAGA group (Experimental): In this arm, patients will undergo PET/CT using 68Ga-NODAGA-LM3 (40ug peptide/150-200MBq) and 68Ga-NODAGA-JR11 (40ug peptide/150-200MBq) on two consecutive days. The scan will be acquired at 1hour post-injection.
  Interventions: Diagnostic Test: 68Ga-NODAGA-LM3 and 68Ga-NODAGA-JR11 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-NODAGA-LM3 and 68Ga-DOTA-LM3 PET/CT — Patients will undergo PET/CT using 68Ga-NODAGA-LM3 (40ug peptide/150-200MBq) and 68Ga-DOTA-LM3 (40ug peptide/150-200MBq) on two consecutive days. The scan will be acquired at 1hour post-injection.
  Arms: LM3 group
Diagnostic Test: 68Ga-NODAGA-LM3 and 68Ga-NODAGA-JR11 PET/CT — Patients will undergo PET/CT using 68Ga-NODAGA-LM3 (40ug peptide/150-200MBq) and 68Ga-NODAGA-JR11 (40ug peptide/150-200MBq) on two consecutive days. The scan will be acquired at 1hour post-injection.
  Arms: NODAGA group

SUMMARY:
Somatostatin receptor antagonists are emerging agents in molecular imaging of neuroendocrine tumors. There're two main antagonist peptides, namely JR11 and LM3, which can be coupled with different chelators, DOTA and NODAGA. Previous studies by our and other groups have revealed the different diagnostic performances of these tracers. However, head-to-head comparison data is still missing. In this study, we aim to evaluate the diagnostic performance of four different antagonists, that is, NODAGA-LM3, DOTA-LM3, and NODAGA-JR11, all labeled with gallium-68.

DETAILED DESCRIPTION:
Patients will be randomly assigned into two arms:

Arm A : 68Ga-NODAGA-LM3 and 68Ga-DOTA-LM3 Arm B : 68Ga-NODAGA-LM3 and 68Ga-NODAGA-JR11

In each arm, patients will undergo PET/CT using assigned tracers. Lesion detection, lesion SUV, and the tumor-to-background ratio will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients of either gender, aged ≥ 18 years.
* Histologically confirmed diagnosis of well-differentiated neuroendocrine tumor.
* A diagnostic computed tomography (CT) or magnetic resonance imaging (MRI) of the tumor region within the previous 6 months prior to dosing day is available.
* At least 1 measurable lesion based on RECIST v1.1.
* Blood test results as follows (White blood cell: ≥ 3*10^9/L, Hemoglobin: ≥ 8.0 g/dL, Platelets: ≥ 50x10^9/L, Alanine aminotransferase / Aspartate aminotransferase / Alkaline phosphatase: ≤ 5 times the upper limit of normal (ULN), Bilirubin: ≤ 3 times ULN)
* Serum creatinine: within normal limits or < 120 μmol/L for patients aged 60 years or older.
* Calculated Glomerular filtration rate (GFR) ≥ 45 mL/min.

Exclusion Criteria:

* Known hypersensitivity to Gallium-68, to NODAGA, to DOTA, to LM3, to JR11 or to any of the excipients of Gallium-68 DOTA-LM3, Gallium-68 NODAGA-LM3, or Gallium-68 NODAGA-JR11.
* Presence of active infection at screening or history of serious infection within the previous 6 weeks.
* Therapeutic use of any somatostatin analog, including long-acting Sandostatin (within 28 days) and short-acting Sandostatin (within 2 days) prior to study imaging. If a patient is on long-acting Sandostatina, then a wash-out phase of 28 days is required before the injection of the study drug. If a patient is on short-acting Sandostatin, then a wash-out phase of 2 days is required before the injection of the study drug.
* Any neuroendocrine tumor-specific treatment between scans.
* Proofs of negative somatostatin receptor expression by previous scans or Immunohistochemical staining results.
* Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide used on such radiopharmaceutical including at any time during the current study.
* Pregnant or breast-feeding women.
* Current history of any malignancy other than neuroendocrine tumor; patients with a secondary tumor in remission of > 5 years can be included.
* Any mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study, and/or evidence of an uncooperative attitude.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Lesion numbers | At 1-hours post-injection
  Determination of lesion numbers of 68Ga-NODAGA-LM3, 68Ga-DOTA-LM3, and 68Ga-NODAGA-JR11 scan.
Standard uptake value (SUV) | At 1-hours post-injection
  Determination of SUV for detected lesions and discernible organs of 68Ga-NODAGA-LM3, 68Ga-DOTA-LM3, and 68Ga-NODAGA-JR11 scan.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjia Zhu, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided